CLINICAL TRIAL: NCT02293460
Title: An International, Multicentre, Efficacy and Safety Study of I10E in Initial and Maintenance Treatment of Patients With Chronic Inflammatory Demyelinating Polyradiculoneuropathy.
Brief Title: Efficacy and Safety Study of I10E in Treatment of Patients With CIDP
Acronym: PRISM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I10E-1302
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Results first posted 2020-03-09 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: Peripheral neuropathy; Disimmune disease; Neurology Chronic disease; Rare disease
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Peripheral Nervous System Diseases; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I10E Arm (Experimental)
  Interventions: Drug: I10E

INTERVENTIONS:
Drug: I10E — Patients who meet all eligibility criteria will receive one dose of IMP at 2g/kg over 2-5 days followed by 7 doses of IMP at 1g/kg over 1-2 day(s), every 3 weeks.
  Duration of treatment period: 21 weeks +/- 7 days.

SUMMARY:
Primary objective:

To assess the efficacy of I10E in improving the disability of patients with CIDP.

Secondary objective:

To assess the safety of I10E in patients with CIDP.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 18 years or more
2. Definite or probable CIDP according to the European Federation of Neurological Societies (EFNS)/Peripheral Nerve Society (PNS) guidelines 2010 clinical and neurophysiological criteria Pure motor CIDP, provided that a diagnosis of multifocal motor neuropathy has been ruled out CIDP associated with monoclonal gammopathy of undetermined significance (MGUS), provided that anti-MAG antibodies titer is lower than the used technique's negativity threshold (1000 BTU for Bühlmann ELISA technique) Lewis-Sumner syndrome
3. Score of at least 2 on the adjusted INCAT disability scale
4. Patient who either :

   1. has never been previously treated with Ig (Ig-naive patient) Or
   2. was previously treated with Ig but is in clinical relapse following treatment withdrawal. In the latter case, the last Ig course shall have been administered no less than 3 months prior to screening

Exclusion Criteria:

1. History of IgA deficiency, unless the absence of anti-IgA antibodies has been documented
2. History of cardiac insufficiency (New York Heart Association [NYHA] III/IV), uncontrolled cardiac arrhythmia, unstable ischemic heart disease, or uncontrolled hypertension
3. History of venous thrombo-embolic disease, myocardial infarction or, cerebrovascular accident
4. Risk factor for blood hyperviscosity such as cryoglobulinemia or haematologic malignancy with monoclonal gammopathy
5. Body mass Index (BMI) ≥40 kg/m²
6. Glomerular filtration rate <80 mL/min/1.73m² measured according to the Modified Diet in Renal Disease (MDRD) calculation
7. Any other ongoing disease that may cause chronic peripheral neuropathy, such as toxin exposure, dietary deficiency, uncontrolled diabetes, hyperthyroidism, cancer, systemic lupus erythematosus or other connective tissue diseases, infection with HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV), Lyme disease, multiple myeloma, Waldenström's macroglobulinaemia, amyloid, and hereditary neuropathy
8. Woman with positive results on a urine pregnancy test or breastfeeding woman or woman of childbearing potential without an effective contraception.
9. Any other serious medical condition that would interfere with the clinical assessment of CIDP or use of I10E or prevent the patient from complying with the protocol requirements
10. Increasing dosage or introduction of a corticotherapy within the last 3 months prior to screening, with oral or systemic corticosteroids at a dose higher than 10 mg daily prednisolone or equivalent. Topical corticosteroids are permitted
11. Treatment within 12 months prior to screening with immunomodulatory or immunosuppressant agents (including but not limited to cyclophosphamide, cyclosporine, interferon-alfa, interferon-beta1a, anti-CD20, alemtuzumab, aziathioprine, etanercept, mycophenolate mofetil, methotrexate and haemopoetic stem cell transplantation)
12. Plasma exchange, blood products or derivatives administered within the last 3 months prior to screening
13. Administration of another investigational product within the last month prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo NOBILE-ORAZIO, MD, Principal Investigator — IRCCS Instituto Clinico Humanitas, Milano, Italy
Locations (33):
- France (7):
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - Hôpital général du CHU de Dijon, Dijon
  - CHU de Nice - Hôpital l'Archet, Nice
  - CHU Paris - Hôpital Pitié salpétrière, Paris
  - Hôpital Pontchaillou, Rennes
  - CHU de saint Etienne - Hôpital nord, Saint-Etienne
  - Hôpital de Hautepierre, Strasbourg
- Italy (7):
  - IRRCS Azienda Ospedaliera Universitaria, Genova
  - IRCCS - Istituto Clinico Humanitas, Milan
  - IRRCS Istituto Nazionale Neurologico Besta, Milan
  - Ospedale San Raffaele IRCCS, Milan
  - Azienda Ospedaliere Universitaria di Padova, Padua
  - Università Cattolica del Sacro Cuore, Roma
  - Azienda Ospedaliere Universitaria san Giovanni, Torino
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Quiron Madrid, Madrid
  - Hospital General Universitario Gregorio, Madrid
  - Hospital clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario i Politècnico La Fe, Valencia
- Tunisia (5):
  - Hôpital Razi, La Manouba, Manouba
  - Hôpital Fattouma Bourguiba, Monastir
  - Hôpital habib Bourguiba, Sfax
  - Hôpital Sahloul, Sousse
  - Hôpital militaire de Tunis, Tunis
- Turkey (Türkiye) (5):
  - Ankara University medical School Neurology, Ankara
  - Hacettepe University Medical School Neurology, Ankara
  - Uludag University Medical School Neurology, Bursa
  - Istanbul UniversityCerrahpasa Medical School Neurology, Istanbul
  - Marmara Universitesi Egitim Ve Arastirma Hastanesi, Istanbul
- United Kingdom (3):
  - St Georges, London
  - Southampton General Hospital, Southampton
  - University Hospital of North Straffordshire, Stratford-upon-Avon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 24 February 2015 and 22 March 2017, 59 subjects from 23 sites signed an informed consent.
Pre-assignment Details: 59 subjects signed an informed consent in the pre-assigment period. Among them, 18 subjects were considered as a screening failure including 3 subjects re-screened and finally enrolled.
  Of 44 enrolled subjects, on subject was discontinued (consent withdrawn by subject) from the study before the first administration of study drug.
Groups:
- Single Arm: This study included patients never previously treated with IgG and patients already treated with IgG but in clinical relapse following IgG therapy discontinuation.
Period: Overall Study
Arm/Group | Single Arm
Started | 43
Completed | 37
Not Completed | 6
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Total Treated Set: All subjects who received at least one infusion of I10E
Arm/Group | Total Treated Set
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 50.0 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  Turkey | 2
  Italy | 16
  United Kingdom | 1
  France | 2
  Tunisia | 8
  Spain | 6
  Poland | 8

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: Responder Rate at End of Study
Description: Responders were defined as patients with a decrease ≥1 point in the adjusted INCAT disability score compared to baseline. Adjusted INCAT disability score can vary from 0 (normal) to 9 (maximal disability).
  If a patient was treated with a not-allowed treatment during the study period, then all adjusted INCAT disability score measured after the intake of these not-allowed treatments were censored.
  If the score at EoS visit was missing, then the Last Observation Carried Forward (LOCF) approach was applied to replace this missing value.
Time Frame: 24 weeks after first treament injection
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Set: All TTS subjects having an available assessment of the primary efficacy criteria.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 42
Participants | 32
Statistical Analysis 1: Comparison: Full Analysis Set; For this single-arm study, the response rate was tested against the historical response rate of 33.3% with a 1-sided Clopper-Pearson exact test at the nominal level of significance of 2.5% on the Full Analysis Set. The null and alternative hypotheses were as follows: H0: pI10E <= 33.3% H1: pI10E > 33.3%; Test type: Superiority — The response rate was tested against the historical response rate of 33.3%; p < 0.0001, exact binomial Clopper-Pearson — One-sided test at nominal level of significance alpha = 2.5 %; Responder rate = 76.2, 95% CI 2-sided [60.5 to 87.9]

ADVERSE EVENTS:
Time Frame: The safety was assessed by recording all AEs occurring during the study, i.e. after signature of the informed consent and until the end of the study recorded (week 24 after inclusion).
Arm/Group | Total Treated Set
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 7/43
Other Adverse Events (participants affected / at risk) | 39/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Treated Set (N=43)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Treated Set (N=43)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Headache (Nervous system disorders) | 20 (79)
Vertigo (Ear and labyrinth disorders) | 3 (5)
Pyrexia (General disorders) | 8 (11)
Asthenia (General disorders) | 4 (4)
Chills (General disorders) | 3 (10)
Malaise (General disorders) | 3 (5)
Nausea (Gastrointestinal disorders) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Influenza (Infections and infestations) | 8 (10)
Urinary tract infection (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT02293460/SAP_002.pdf
  • Study Protocol (2017-05-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT02293460/Prot_003.pdf